CLINICAL TRIAL: NCT05670158
Title: Study on the Inner Ear Immunisation Post-cohlear Implantation and Perilymph Molecular Profiling in Sensorineural Hearing Loss
Brief Title: Immunity After Cochlear Implantation and Perilymph Molecular Profiles in Sensorineural Hearing Loss
Acronym: PERILOTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0380
Record Dates: First submitted 2022-12-12; First posted 2023-01-04 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sensorineural Hearing Loss
Keywords: Perilymph; Proteomics; Metabolomics; Sensorineural hearing loss; Residual hearing; Cochlear implantation
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study will recruit individuals eligible for cochlear implantation surgery. In parallel, the control group will be formed from normal hearing patients - candidates for other otological interventions. The two groups will be matched by age and gender of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Cochlear Implantation" group (Experimental): 50 patients with sensorineural hearing loss eligible for cochlear implantation surgery. The blood and perilymph sampling will be performed during surgery (visit V1). The blood sampling will be additionally done during the visits V2, V3 and V4. After the visit V4, this arm will be subdivided into 2 groups: group 1, 15 patients with the delayed residual hearing loss, and group 2,15 patients with preserved residual hearing. For these 30 patients, blood sampling will be also performed during the visit V5.
  Interventions: Biological: Blood sampling; Procedure: Perilymph sampling
- Control group (Other): 30 normally hearing patients who will undergo through an otological surgery other than cochlear implantation. A blood sampling will be performed during surgery (visit V1) as well as during the visits V2 and V3.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood will be collected into 2 EDTA and 1 heparin tube. The 2 EDTA tubes (4ml of blood in each) will be transported on ice to the proteomics platform in the next three hours, centrifuged and stored on -80 degrees Celcius in low-binding tubes for further molecular analysis. 1 heparin tube (5mL) will be sent to the Bacteriology-Virology Department for the active PBMC counting.
Procedure: Perilymph sampling — The perilymph collection will be performed during the cochlear implantation surgery at the same time as the round window opening. 5 to 15 microliters will be aspirated using an atraumatic spinal needle mounted onto 1 ml insulin syringe.
  Arms: "Cochlear Implantation" group

SUMMARY:
Many patients receiving cochlear implant (CI) have some residual hearing prior to implantation surgery. However, approximately one third of them will lose it in next 6 months after cochlear implantation. Although the mechanisms involved in the residual audition loss remain unknown, animal experiments suggest the role of inflammatory or immune reaction in the cochlea. The goal of this project is to search in the perilymph (a fluid which fills the scala vestibuli and scala tympani of the cochlea) some predictive biomarkers of the residual hearing loss using modern proteomics and immunological techniques. A parallel search for blood biomarkers of post-implantation residual hearing loss and for molecular and cellular evidences of immune response to cochlear implantation will be performed.

The study will recruit 50 subjects-candidates for cochlear implantation surgery; 30 normally hearing individuals eligible for other types of otological interventions will form a control group. For all the participants blood samples will be collected and preserved. In addition, the perilymph sampling will be performed during cochlear implantation surgery.

This project relies on the calculation that from 50 patients post-cochlear implantation, 15 patients will form a group with maintained residual hearing and 15 will display delayed hearing loss. For these 30 subjects together with the control group the blood biomarkers search will be performed.

For the group of implanted patients, the follow-up will last for 12 months with 6 visits in total :

* the inclusion visit V0 during which the study will be presented and the consent form will be signed
* the surgery visit V1 with blood sample and perilymph collection
* the activation visit V2, 1 month ± 1 week after V1, visit V3 3 months ± 7 days after V1, V4 6 months ± 7 days after V1, V5 12 months ± 1 month after V1. During each of this visit blood sampling will be performed.

For the control group, the follow up will be 6 months long with 4 visits in total arranged during the routine follow-up appointments:

* the inclusion visit V0 during which the study will be presented and the consent form will be signed
* the surgery visit V1, the 1 month visit V2 and the 6 months visit V3 during which the blood sampling will be performed.

DETAILED DESCRIPTION:
With the progress of technologies and surgical methods, cochlear implantation, initially proposed only to patients with completely non-functional inner ear, can be now performed on individuals with still some measurable hearing left in some frequencies. Such patients can additionally benefit from a special treatment by electric-acoustic stimulation (EAS). Combining the electric stimulation with cochlear implant (CI) and acoustic amplification of residual hearing using a conventional hearing aid (HA) can drastically improve one's quality of life and ameliorate the performance in noisy environment as well as music perception.

Since the main condition for EAS is the residual hearing preservation, it is important to understand the reasons of its loss post-cochlear implantation. This loss can occur in 2 periods:

* Early after surgery (˂ 1 month): mainly due to the trauma from electrode insertion. This risk decreases with the development of surgical techniques. Another possible reason is early inflammation processes in the cochleae.
* Later after surgery (˃ 1 month): occurs mainly about 3 months post-implantation in 30-40 % of patients. This loss is the main reason for dropping out the EAS leaving the patient to rely on CI only.

Animal studies suggest that the delayed residual hearing loss might happen as consequence of cochlear fibrosis development, supposedly due to the inflammation and foreign body response to the CI materials within the cochlea. In its natural state, the cochlea does not contain any immune cells and is well protected from immune stimulation by infectious agents. Cochlear implantation, however, provides a single clinical cause for infectious or autoimmune fibrosis. Such immune response might be provoked by autoantigens against cochlear proteins like Cochline or TectB. This study aims to search blood markers of immunisation against inner ear proteins after cochlear implantation. Another goal is to seek potential biomarkers of delayed residual hearing loss directly in perilymph. Proteomic analysis will be performed using Liquid Chromatography - High Resolution Mass Spectroscopy (HRMS) technique.

The main objective of this study is

* to identify, in the perilymph of implanted patients, biomarkers predictive of the delayed residual hearing loss
* to identify blood biomarkers predictive of delayed residual hearing loss in implanted patients

The secondary objectives are

* to describe qualitatively and quantitatively the time evolution for blood biomarkers of interest after cochlear implantation
* to correlate quantitative values of identified biomarkers with clinical data of implanted patients
* to identify perilymph and blood biomarkers of early residual hearing loss post-cochlear implantation
* depending on molecular profiles identified, to study metabolic pathways and mechanisms involved in delayed residual hearing loss post-cochlear implantation
* to seek for blood indicators in favour of anti-cochlear immunisation through screening for peripheral blood mononuclear cells (PBMC)
* to create a bio collection of human perilymph and blood serum biobank of cochlear implants users for future proteomics/molecular studies

ELIGIBILITY:
Inclusion Criteria for the "Cochlear implantation" group :

* Patients aged 18 years or more
* Indication for the cochlear implantation surgery according to the criteria of French National Authority for Health (Severe to profound sensorineural deafness with indication for cochlear implant surgery: Intelligibility less than or equal to 50% when performing vocal audiometry tests with Fournier's list in free field with recent devices.)
* Presence of "useful" residual hearing ≤ 80 dB on at least 2 consecutive frequencies (in air conduction) from the range 125, 250, 500, 1000 kHz on pure-tone audiometry
* Patients given their free and informed written consent
* Patients affiliated to a French social security system

Inclusion Criteria for the "Control" group:

* Patients aged 18 years or more
* Indication for otological surgery of the middle ear (excluding active infectious or inflammatory pathology e.g. myringoplasty, ossiculoplasty, cure for otosclerosis)
* Normal hearing (non affected inner ear): average hearing loss (mean threshold for the frequencies 500, 1000, 2000, 4000 Hz) ≤ 35 dB in bone conduction
* Patients given their free and informed written consent
* Patients affiliated to a French social security system

Exclusion Criteria for the "Cochlear implantation" group:

* Contraindication to surgery detected during the preoperative assessment
* Pre-implantation cochlear assessment unfavorable to the implantation surgery
* Absence of residual hearing shown by preoperative audiometry
* History of bacterial labyrinthitis or bacterial meningitis
* Cochlear ossification shown on preoperative imaging
* Homozygous pathogenic mutations identified by molecular diagnosis of the SCL26A5 (prestin), TECTB (Beta-Tectorin) genes, and heterozygous of the COCH gene (Cochlin) prior to implantation (if available)
* Vulnerable subject: minors, protected adults as defined by the Public Health Code, pregnant or breastfeeding women, subject under guardianship or subject deprived of liberty
* Participation in another pharmacological therapeutic interventional clinical research

Exclusion Criteria for the Control group:

* Contraindication to surgery detected during the preoperative assessment
* Fluctuating hearing = fluctuating hearing thresholds on at least one ear (shown by past bone conduction pure-tone audiometries)
* History of bacterial labyrinthitis or bacterial meningitis
* Middle ear infection or inflammation on the day of the surgery
* Chronical immune or inflammatory disease
* Active viral or bacterial infection on the day of inclusion visit or surgery
* Fever on the day of the first blood sample
* Vulnerable subject: minors, protected adults as defined by the Public Health Code, pregnant or breastfeeding women, subject under guardianship or subject deprived of liberty
* Participation in another pharmacological therapeutic interventional clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Expression levels of proteins and metabolites in the perilymph before surgery in the 2 groups of implanted patients | Before cochlear implantation surgery (V1)
  Expression levels of proteins and metabolites identified by high-resolution mass spectrometry (Lc-HRMS) in the perilymph of group 1, "delayed residual hearing loss" and group 2, "maintained residual hearing" patients, collected before cochlear implantation surgery
Expression levels of proteins and metabolites in the blood before surgery in the 2 groups of implanted patients | Before cochlear implantation surgery (V1)
  Expression levels of proteins and metabolites identified by high-resolution mass spectrometry (Lc-HRMS) in the blood of group 1 "delayed residual hearing loss" and group 2 "maintained residual hearing" patients, collected before cochlear implantation surgery

SECONDARY OUTCOMES:
PBMC cell counting | Before cochlear implantation surgery (V1)
  Counting of activated blood immune cells, using FACS technique after the PBMC cells culture is performed
PBMC cell counting | At 1 month post-implantation (V2)
  Counting of activated blood immune cells, using FACS technique after the PBMC cells culture is performed
PBMC cell counting | At 3 months post-implantation (V3)
  Counting of activated blood immune cells, using FACS technique after the PBMC cells culture is performed
PBMC cell counting | At 6 months post-implantation (V4)
  Counting of activated blood immune cells, using FACS technique after the PBMC cells culture is performed
PBMC cell counting | At 12 months post-implantation (V5)
  Counting of activated blood immune cells, using FACS technique after the PBMC cells culture is performed
Expression levels of identified molecules in the 2 groups of implanted patients after the surgery | At 1 month post-implantation (V2)
  Expression levels of identified molecules for each group over time
Expression levels of identified molecules in the 2 groups of implanted patients after the surgery | At 3 months post-implantation (V3)
  Expression levels of identified molecules for each group over time
Expression levels of identified molecules in the 2 groups of implanted patients after the surgery | At 6 months post-implantation (V4)
  Expression levels of identified molecules for each group over time
Expression levels of identified molecules in the 2 groups of implanted patients after the surgery | At 12 months post-implantation (V5)
  Expression levels of identified molecules for each group over time

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No